CLINICAL TRIAL: NCT03877705
Title: Effect of Dissolving Xylitol Chewable Tablets Versus Xylitol Chewing Gum on Salivary pH and Bacterial Count in Geriatric Bedridden Patients : Randomized Clinical Trial
Brief Title: Xylitol Chewable Tablets Versus Xylitol Chewing Gum in Geriatric Bedridden Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Manar abd elmageed ahmed, Manar abd El mageed ahmed, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Xylitol tabs vs xylitol gum
Record Dates: First submitted 2019-03-12; First posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Saliva Altered; Plaque
Keywords: Dental Plaque , salivary pH
MeSH Terms: conditions — Plaque, Amyloid; Dental Plaque

STUDY DESIGN:
Intervention Model Description: Geriatric bedridden patients
Who Masked: Investigator, Outcomes Assessor
Masking Description: The operator will be blinded to material and assessors will be blinded to the material assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dissolving xylitol chewable tablets (Experimental): Listerine ready tabs 3 times/day
  Interventions: Drug: Listerine ready tabs
- Xylitol chewing gum (Active Comparator): Trident original 3 times/day
  Interventions: Drug: Listerine ready tabs

INTERVENTIONS:
Drug: Listerine ready tabs — Technically, it's a rectangular-shaped, bilayer-compressed tablet that once chewed, creates just enough liquid to swish around your mouth to get a whole-mouth clean feeling.As manufacture claimed the tablet is easy to use just in three simple steps: chew (to activate), swish (to clean), then swallow as unlike mouthwashes which may contain alcohol and other ingredients not intended for ingestion, Listerine Ready Tabs are alcohol-free and safe to swallow which is highly suitable for bedridden patients.
  Other Names: Listerine chewable tablets

SUMMARY:
This study will be conducted to evaluate the effectiveness of using dissolving Xylitol chewable tablets versus xylitol chewing gum with bedridden geriatric patients in increasing salivary pH and decreasing bacterial count in both saliva and interdental plaque.

DETAILED DESCRIPTION:
This study will be conducted to evaluate the value of using dissolving Xylitol chewable tablets versus xylitol chewing gum with bedridden geriatric patients ,as an alternative to tooth brushing and mouth rinsing, in increasing salivary pH and decreasing bacterial count in both saliva and interdental plaque.plaque and salivary sampling will be taken in certain time ,at baseline T0, then after 5minutes T1, then at 15 days T3. Salivary pH will be measured by using pH meter and streptococcus mutans bacterial count will be calculated through culture in mitis salivarius bacitracin

ELIGIBILITY:
Inclusion Criteria:

1. Age range above 65 years old
2. Bedridden patients
3. Males or females
4. Concious patients
5. Co-operative patients approving to participate in the trial.
6. Subjects who signed informed consent

Exclusion Criteria:

1. Individuals had taken antibiotics during the last four weeks or anticipated doing so during the study
2. Subjects who wore removable prosthesis
3. Patients with systemic diseases that have any oral manifestations
4. History of Smoking
5. Allergy to any of chewing gum or tablets ingredients
6. Evidence of tempromandibular joint disorders
7. Presence of intraoral infections
8. Currently using any mouth rinse

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Salivary bacterial count | 15 days
  Streptococcus mutans count in saliva

SECONDARY OUTCOMES:
Interdental plaque Bacterial count | 15 days
  Mesial and distal Interdental plaquns streptococcus mutans count

OTHER OUTCOMES:
Salivary pH | 15 days
  Degree of acidity or alkalinity of salivary pH

CONTACTS AND LOCATIONS:
Overall Officials: Faculty Of Dentistry, Faculty, Study Director — Cairo University
Locations (1):
- Faculty of dentistry, Al Manyal, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
A paper of the research will be published internationally after results calculation

REFERENCES:
- [Background] Oza S, Patel K, Bhosale S, Mitra R, Gupta R, Choudhary D. To Determine the Effect of Chewing Gum Containing Xylitol and Sorbitol on Mutans Streptococci and Lactobacilli Count in Saliva, Plaque, and Gingival Health and to Compare the Efficacy of Chewing Gums. J Int Soc Prev Community Dent. 2018 Jul-Aug;8(4):354-360. doi: 10.4103/jispcd.JISPCD_54_18. Epub 2018 Jul 18. PMID 30123770
- See also: Free PMC article — https://www.ncbi.nlm.nih.gov/m/pubmed/30123770/
- Available data/document: Individual Participant Data Set: Pubmed — http://www.ncbi.nlm.nih.gov/m/pubmed/30455769/?i=6&from=xylitol%20review

DOCUMENTS (1):
  • Study Protocol (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT03877705/Prot_000.pdf